CLINICAL TRIAL: NCT01418963
Title: A Single- and Multiple Ascending-Dose, Randomized, Double-Blind, Placebo-Controlled Study in Two Single-Center Study Parts to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO5285119 Following Oral Administration in Healthy Subjects
Brief Title: A Study of RO5285119 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP25694
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active (Experimental)
  Interventions: Drug: RO5285119
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RO5285119 — single and multiple ascending oral doses
  Arms: Active
Drug: placebo — single and multiple oral doses
  Arms: Placebo

SUMMARY:
This two-part, randomized, double-blind, placebo-controlled study will assess the safety, pharmacokinetics and pharmacodynamics of single and multiple ascending oral doses of RO5285119 in healthy volunteers. Anticipated time on study will be up to 9 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults, 18 to 45 years of age (Part 1) or healthy male or female adults, 18 to 65 years of age (Part 2)
* Body mass index (BMI) 18.0 to 30.0 kg/m2 inclusive
* Female subjects must be surgically sterile or postmenopausal
* Male subjects must use a barrier method of contraception for the duration of the study and for the three months after the last dosing

Exclusion Criteria:

* History or presence of any significant disease or disorder
* Positive for hepatitis B. hepatitis C or HIV infection
* History of drug or alcohol abuse or suspicion of regular consumption of drugs of abuse
* Participation in an investigational drug or device study within 3 months prior to first dosing
* Donation of blood within 3 months prior to first dosing
* Regular smoker (>5 cigarettes, >3 pipe-fulls, >3 cigars per day)
* History of hypersensitivity or allergic reactions
* Part 2: Contraindications for MRI scans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to 5 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration - time curve (AUC) | up to 5 weeks
Pharmacodynamics (neurological effects): Profile of Mood States/Bond&Lader VAS/smell test/C-SSRS | up to 5 weeks
Pharmacodynamics: Biomarker levels (ACTH, prolactin, cortisol, vasopressin) | up to 5 weeks
Pharmacodynamics: Functional Magnetic Resonance Imaging | up to 5 weeks
Food effect: Comparison of single dose pharmacokinetics (AUC) in fasted and fed state (Part 1b) | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- France (2):
  - Rennes
  - Strasbourg

REFERENCES:
- [Derived] Derks M, Lennon-Chrimes S, Guenther A, Squassante L, Wandel C, Szczesny P, Paehler A, Kletzl H. Bioavailability and pharmacokinetic profile of balovaptan, a selective, brain-penetrant vasopressin 1a receptor antagonist, in healthy volunteers. Expert Opin Investig Drugs. 2021 Aug;30(8):893-901. doi: 10.1080/13543784.2021.1948009. Epub 2021 Jul 16. PMID 34176392